CLINICAL TRIAL: NCT06816654
Title: Retrospective Evaluation of the Impact of Epidural on the Risk of Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head of Clinical Trial Unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-PERIHPeriPartum
Record Dates: First submitted 2025-01-31; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Epidural anesthesia; Postpartum hemorrhage; Obstetric analgesia; Neuraxial anesthesia; Instrumental delivery; Obstetrical trauma
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vaginal deliveries: Patients who gave birth vaginally at Brugmann University Hospital between January 1, 2020 and December 31, 2021.
  Interventions: Other: Data extraction from medical records

INTERVENTIONS:
Other: Data extraction from medical records — Data extraction from medical records

SUMMARY:
Postpartum hemorrhage (PPH) is a major complication of childbirth. Epidurals are often implicated in the onset of postpartum hemorrhages. Given the paradoxical data in the literature, the investigators wished to retrospectively evaluate the impact of epidurals on the risk of PPH, instrumental delivery and the occurrence of PPH risk factors.

The investigators retrospectively analyzed 5753 records of patients who gave birth vaginally at Brugmann University Hospital between January 1, 2020 and December 31, 2021. The primary objective was to assess whether epidurals pose a risk of postpartum hemorrhage. Secondly, the investigators assessed whether epidurals pose a greater risk of instrumentation of delivery and emergence of PPH risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who gave birth vaginally at the Brugmann University Hospital Horta site between January 1, 2020 and December 31, 2021.

Exclusion Criteria:

* Patients who gave birth before 25 weeks.
* Patients who gave birth outside of hospital.
* Patients who had recourse to a medical termination of pregnancy (MTP).
* Patients who gave birth by cesarean section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who gave birth vaginally at the Brugmann University Hospital Horta site between January 1, 2020 and December 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 5753 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Postpartum blood loss | Up to 24 hours after the birth of the baby
  Total blood loss is analyzed according to a standardized protocol: use of the calibrated field of the collection bag and of a precision scale to weigh the blood soaked compresses

SECONDARY OUTCOMES:
PPH risk factors | Data extraction in medical files from January 1st 2020 till December 31th 2021
  Presence/absence of one or more PPH risk factors (yes/no) such as : uterine atony, placental abnormalities, obstetric trauma, and coagulopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Botti, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No